CLINICAL TRIAL: NCT05821725
Title: Clinical Study to Evaluate the Effects of a Topical Hyaluronic Acid (HA) Gel on Postoperative Pain and Wound Healing at Palatal Donor Sites in Subjects Undergoing Mucogingival Procedures
Brief Title: Effects of Topical Hyaluronic Acid Gel on Postoperative Pain and Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRO-2022-09-WH-BZ-ZM
Record Dates: First submitted 2023-03-22; First posted 2023-04-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2023-08

CONDITIONS: Palatal Wound
Keywords: Topical hyaluronic acid; Postoperative pain; Wound healing; Epithelialized; Palate; supportive care; Treatment; Prevention
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): A gel containing Hyaluronic acid in combination with a hemostatic sponge
  Interventions: Device: Hyaluronic acid
- Group II (Active Comparator): A hemostatic sponge alone
  Interventions: Device: Control

INTERVENTIONS:
Device: Hyaluronic acid — Hyaluronic acid and hemostatic sponge
  Arms: Group I
Device: Control — Hemostatic sponge
  Arms: Group II

SUMMARY:
This clinical study aims to investigate the impact of a topical hyaluronic acid (HA) gel on postoperative pain and wound healing at palatal donor sites in patients undergoing mucogingival procedures involving a de-epithelialized gingival graft (DGG) from the palate. The study design is a Phase III, randomized, double-blind, parallel-group, clinical trial, conducted in a single center, with 30 subjects aged 18-70 years.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18-70 years of age
* Informed Consent Form signed and availability for the duration of the study
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study
* Clinical indication for mucogingival surgery that requires a de-epithelialized gingival graft (DGG) from the palate
* Willingness to provide information related to their medical history
* Minimum of 10 uncrowned permanent natural teeth (excluding third molars)
* Normal salivary flow

Exclusion Criteria:

* Oral pathology, chronic disease, or a history of allergy to testing products
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study
* Subject participating in any other clinical study
* Subject pregnant or breastfeeding
* Subject allergic to oral care products, personal care consumer products, or their ingredients
* Extended use of antibiotics or therapeutic mouthwash any time during the three months prior to entry into the study
* A medical history reporting that the subject has a current systemic or autoimmune disease, such as diabetes, lupus, etc
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Wound healing area | Baseline
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter
Wound healing area | 3 days after surgery
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter
Wound healing area | 7 days after surgery
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter
Wound healing area | 14 days after surgery
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter
Wound healing area | 21 days after surgery
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter
Wound healing area | 42 days after surgery
  Wound size will be assessed at Baseline after obtaining the graft, and 3, 7, 14, 21, and 42 days after surgery via direct measurement with a Periodontal Probe UNC 15 (Hu-Friedy, United States), length and height of the wound will be measured and recorded to the nearest millimeter

SECONDARY OUTCOMES:
Pain assessment | Baseline
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.
Pain assessment | 3 days after surgery
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.
Pain assessment | 7 days after surgery
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.
Pain assessment | 14 days after surgery
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.
Pain assessment | 21 days after surgery
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.
Pain assessment | 42 days after surgery
  Pain will be assessed via Visual Analog Scale (VAS) at Baseline, 3, 7, 14, 21, and 42 days after surgery. A line of 10 cm will be used in which at the left end of the line will have a verbal anchor stating "No pain" and on the other end the verbal anchor of "The most intense pain that I ever felt". The subjects will place a mark on the line and the distance from the beginning of the line up to the mark will be measured and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faveri, DDS, PhD, Study Director — Faveri Academy
Locations (1):
- Faveri Academy, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No